CLINICAL TRIAL: NCT07059299
Title: NeoTISLEGA - A Phase Ib Trial Evaluating the Safety and Activity of Neoadjuvant Combination of Tislelizumab Plus FLOT for Resectable Esophagogastric Adenocarcinoma
Brief Title: A Phase Ib Trial Evaluating the Safety and Activity of Neoadjuvant Combination of Tislelizumab Plus FLOT for Resectable Esophagogastric Adenocarcinoma
Acronym: NeoTISLEGA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: BeiGene (Industry); Universitätsklinikum Leipzig (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCL-IKF-NeoTISLEGA; 2024-519993-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-03; First posted 2025-07-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Esophagogastric Junction Adenocarcinoma; Gastric Adenocarcinoma; Esophageal Adenocarcinoma; Resectable Esophagogastric Adenocarcinoma; Neoadjuvant Therapy
Keywords: gastric cancer; FLOT; Tislelizumab; neoadjuvant
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose intensification (Level 1 and 2) (Experimental): In the dose intensification part of the trial, eligible patients will be enrolled in a staggered approach with 6 patients for each successive dose level:
  Dose level 1 (n=6):
  * 4 cycles tislelizumab (200 mg, i.v. on day 1 Q3W ) plus
  * 6 cycles: FLOT (docetaxel 50 mg/m², oxaliplatin 85 mg/m², leucovorin 200 mg/m² and 5-FU (5-fluorouracil) 2600 mg/m², all i.v. on day 1 Q2W)
  Dose level 2 (n=6):
  * 5 cycles tislelizumab (200 mg, i.v. on day 1 Q3W) plus
  * 8 cycles: FLOT (docetaxel 50 mg/m², oxaliplatin 85 mg/m², leucovorin 200 mg/m² and 5-FU 2600 mg/m², all i.v. on day 1 Q2W)
  The maximum dose level at which one or less out of 6 patients experienced a DLT is considered an optimal dose.
  In the expansion part of the trial, the dose level classified as optimal dose will be extended by a further 6 patients (12 patients in total for the optimal dose level).
  Interventions: Drug: Tislelizumab; Drug: FLOT Chemotherapy

INTERVENTIONS:
Drug: Tislelizumab — humanized immunoglobulin G4 (IgG4)-variant monoclonal antibody (mAb) against human programmed cell death-1 (PD-1)
Drug: FLOT Chemotherapy — docetaxel 50 mg/m², oxaliplatin 85 mg/m², leucovorin 200 mg/m² and 5-FU 2600 mg/m², all i.v. on day 1 Q2W

SUMMARY:
With this trial, we aim to evaluate a new combination therapy with tislelizumab and FLOT chemotherapy before surgery (neoadjuvant) for locally advanced, resectable adenocarcinoma of the esophagus or stomach (EGA). The aim of this phase Ib trial is to determine whether this combination is safe and clinically active enough to support the continuation of this concept in subsequent trials investigating novel drug combinations in the neoadjuvant setting of locally advanced EGA. As many patients are unable to tolerate the postoperative part of the standard therapy concept, we aim here to assess a prolongation of preoperative therapy to 6 or 8 applications of FLOT, instead of the routinely administered 4 pre- and 4 postoperative applications, in combination with tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* has given written informed consent.
2. Patient is ≥ 18 years of age at time of signing the written informed consent.
3. Patient has histologically proven locally advanced (cT2-4 , any cN , M0 OR any cT, cN+, M0 stage) gastric, esophageal or esophagogastric junction adenocarcinoma that:

   1. Is considered technically resectable.
   2. Does not involve distant site of the peritoneal cavity.

      * confirmed by diagnostic laparoscopy for all patients with tumors located in the stomach and those with type 2 and 3 GEJ adenocarcinomas according to ESMO guideline recommendation [Lordick et al. 2022].
      * Type 1 GEJ and esophageal adenocarcinomas can be enrolled without diagnostic laparoscopy (which is in line with guidelines and the current routine practice in Germany).
4. Tumor material is available for local assessment of PD-L1 (CPS) and dMMR/MSI-status at the investigator´s site.
5. Patient has an ECOG performance status 0 or 1.
6. Patients has adequate blood count, liver-enzymes, and renal function:

   1. ANC (Absolute neutrophil count) > 1,500 cells/μL without the use of hematopoietic growth factors.
   2. Platelet count ≥ 100 x 10^9/L (>100,000 per mm3).
   3. Hemoglobin ≥ 9 g/dL.
   4. Serum total bilirubin ≤ 1.5x institutional upper normal limit (ULN).
   5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN.
   6. Patients not receiving therapeutic anticoagulation must have an INR ≤ 1.5 ULN and aPTT ≤ 1.5 ULN. The use of full dose anticoagulants is allowed (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of inclusion.
   7. Serum Creatinine ≤ 1.5 x ULN and a calculated creatinine clearance rate ≥ 50 mL /min.
7. Female patients defined as women of childbearing potential (WOCBP) must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for 4 months after last dose of tislelizumab or 6 months after the last dose of chemotherapy, whatever is later. Male patients with WOCBP partners must agree to remain abstinent (refrain from heterosexual intercourse) or use barrier contraceptives during the above period. Furthermore, male patients must refrain from donating sperm during this same period.

   * There are no data that indicate special gender distribution. Therefore, patients will be enrolled gender-independently in this trial.

Exclusion Criteria:

1. Patient received previous (radio)chemotherapy or immunotherapy for the same condition or within the past five years for any other cancerous condition.
2. Patient received prior partial or complete esophagogastric resection.
3. Patient has known hypersensitivity to any component of the tislelizumab formulation as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein and/or any known contraindication (including hypersensitivity) to one of the study drugs.
4. Patient has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
5. Patient has lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within three months of the study randomization, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.).
6. Patient has inadequate cardiac function (LVEF value < 50 %) as determined by echocardiography.
7. Patient has a known complete absence of dihydropyrimidine dehydrogenase (DPD) activity.
8. Patient received treatment with brivudine, sorivudine or their chemically related analogues within 28 days prior to study enrollment.
9. Patients has pernicious anemia or other megaloblastic anemia due to vitamin B12 deficiency.
10. Patient has peripheral sensitive neuropathy with functional deficits.
11. Patient has a medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF; New York Heart Association Class II to IV). Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any MI related symptoms should have a cardiologic consultation during screening to rule out MI.
12. Patient has a corrected QT interval (QTc) prolongation to > 470 ms (females) or >450 ms (males) based on average of the screening triplicate12-lead ECG.
13. Participant has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
14. Patient has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
15. Patient has active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C (HBV/HCV) infection. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA. Subjects with past or resolved HBV infection are eligible only if they meet all of the following criteria:

    * HBsAg(-) (for > 6 months off anti-viral treatment)
    * Anti-HBc(+) (IgG or total Ig)
    * HBV DNA undetectable
    * Absence of cirrhosis or fibrosis on prior imaging or biopsy
    * Absence of HCV co-infection or history of HCV co-infection
    * Access to a local hepatologist during and after the study
16. Patient has active or history of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
17. Patient received treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within four weeks or five half-lives of the drug, whichever is longer, prior to study enrollment.
18. Patient received treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to study enrollment. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
19. Patient received prior allogeneic bone marrow transplantation or prior solid organ transplantation.
20. Patient received live, attenuated vaccine within 30 days prior initiation of study drug.
21. Patient has any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
22. Patient participated in another interventional clinical study according to Medicines Act within 28 days prior to study enrollment or participation in a clinical study according to Medicines Act at the same time as this study unless it is an observational / non-interventional study or during the follow-up period of an interventional study.
23. Patient has taken an investigational drug within 28 days prior to initiation of study drug.
24. Female patients, who are pregnant or breast feeding or planning to become pregnant within 7 months after the last dose of study treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility rate | up to 8 months
  Feasibility rate, defined as proportion of patients receiving the protocol treatment before surgery ('neoadjuvant') according to the planned schedule without occurrence of at least one dose-limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, Prof. Dr., Principal Investigator — Universitätsklinikum Leipzig; Salah Eddin Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (4):
- Germany (4):
  - Krankenhaus Nordwest GmbH Institut für Klinisch-Onkologische Forschung (IKF), Frankfurt
  - Hämatologisch-Onkologische Praxis Eppendorf (hope), Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar München der TU München, München